CLINICAL TRIAL: NCT03493971
Title: Impact of Carotid Endarterectomy and Stenting on Hemodynamics, Fluid-structure Interaction, Autonomic Modulation, and Cognitive Brain Function
Brief Title: Hemodynamics and Autonomic and Cognitive Performance After Carotid Revascularization Procedures
Acronym: BAROX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Collaborators: Emory University (Other); University of Pavia (Other)
Responsible Party: Principal Investigator, Massimiliano M. Marrocco-Trischitta, MD, PhD, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62/int/2017; PE-2013-02355484 (Other Grant/Funding Number: Ministero della Salute, Italia)
Record Dates: First submitted 2017-12-05; First posted 2018-04-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Carotid Artery Diseases
Keywords: carotid endarterectomy; carotid stenting; autonomic function; computational fluid dynamic; cognitive function
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotid artery stenting (CAS) (Active Comparator): Carotid revascularization performed using CAS
  Interventions: Procedure: Carotid revascularization performed using CAS
- Carotid endarterectomy (CEA) (Active Comparator): Carotid revascularization performed using CEA
  Interventions: Procedure: Carotid revascularization performed using CEA

INTERVENTIONS:
Procedure: Carotid revascularization performed using CAS — Carotid artery stenting (CAS) is an endovascular stent procedure used to treat narrowing of the carotid artery and decrease the risk of stroke
  Arms: Carotid artery stenting (CAS)
Procedure: Carotid revascularization performed using CEA — Carotid endarterectomy (CEA) is a surgical procedure used to correct stenosis in the common carotid artery or internal carotid artery and reduce the risk of stroke
  Arms: Carotid endarterectomy (CEA)

SUMMARY:
Carotid revascularization procedures are performed for more than 87% of cases in patients with asymptomatic internal carotid stenosis (ICS), who are assumed to have a life expectancy of at least 5 years. Hence, the investigators aim to compare carotid artery stenting (CAS) with carotid endarterectomy (CEA) in terms of long-term prognostic endpoints in patients with uneventful perioperative course. CEA and CAS, as a consequence of either surgical trauma or mechanical stimuli related to the compliance mismatch between the stented segment and the native artery, may perturb carotid baroreceptors function causing an impairment of cardiovascular autonomic control. Also, CEA and CAS result in different postoperative geometric features of carotid arteries that entail relevant modifications of rheological parameters, that may be associated with the risk of local complications. Finally, long-term and sustained cognitive benefits after CAS as compared to CEA are yet to be demonstrated.

DETAILED DESCRIPTION:
Hypothesis and Significance: Late clinical outcome and prognosis after CAS may be inferior to that after CEA in terms of autonomic modulation, hemodynamic remodeling, and cognitive function.

Specific Aim: 1) To compare the impact of CEA and CAS on long-term post-operative baroreceptor function and on cognitive brain function, and analyze their influence on clinical outcome. The specific goal is to assess the potential correlation between post-operative autonomic and cognitive function. 2) To assess the solicitation on the carotid wall due to CAS as compared to CEA through structural analysis and mechanical modeling. The specific goal is to assess the potential correlation between stenting, wall damage, baroceptor impairment, and late neurological sequelae. 3) To assess the post-operative carotid hemodynamics combining medical image analysis, clinical data, and computer simulations. The specific goal aims at correlating both local (e.g., wall stress stress) and global phenomena (controlateral flow, arterial stiffening) with baroreflex function and post-operative neurological outcomes.

Experimental Design Aim 1: A computerized method requiring small operator interaction will be used to assess indices of autonomic sympathovagal balance directed to the sinoatrial node, sympathetic vasomotor modulation, and baroreflex gain, all from spontaneous beat-by-beat variations of the R-R interval and systolic arterial pressure (SAP) variability, considering only sinus rhythm conditions. After electrode and sensor positioning, patients will be maintained for 10 minute in resting supine position, necessary for stabilization, subsequently blood pressure waveforms, electrocardiogram and respiratory activity will be continuously recorded during a nominal 5-minute baseline and then for subsequent 5-minute period of active standing.

Cardiovascular signals will be acquired by a 4 channel digital polygraph. The electrocardiogram will be recorded with two electrodes placed on the patient's chest, breathing pattern will be recorded by a piezoelectric belt and finger arterial blood pressure will be continuously monitored by a CNAP 500 HD continuous noninvasive hemodynamics monitor (CNSystems Medizintechnik AG, Austria). As described previously, (8) a series of indexes indirectly reflecting autonomic cardiovascular modulation will be derived from the spectral analysis of R-R interval and SAP variability. Postoperative cardiovascular autonomic control will be correlated to clinical outcome and measures of cognitive performance. Enrolled patients will be submitted to Mini-Mental State Examination for general cognitive impairment screening. Cognitive P300 evoked potentials will be then recorded, before and after treatment, with Ag/AgCl electrodes with a Brain Vision Recorder (Brain Products GmbH, Gilching, Germany). P300 evoked potentials will be generated after a binaurally presented tone discrimination paradigm (odd-ball paradigm) with frequent (80%) tones of 1000 Hz and rare (20%) target tones of 2000 Hz at 75 dB HL. Filter bandpass will be 0.01 to 30 Hz. Active electrodes will be placed at Cz (vertex) and Fz (frontal), respectively, and referenced to linked earlobe A1/2 electrodes (10/20 international system). During the paradigm, the patients will be instructed to keep a running mental count of the rare 2000-Hz target tones. To verify attention, P300 recordings with a discrepancy of>10% between the actual number of stimuli and the number counted by the patients will be rejected and repeated. P300 evoked potential recording will result in a stable sequence of positive and negative peaks. Latencies in milliseconds (ms) of the cognitive P300 peak will be assessed. To confirm reproducibility, two sets of P300 measurements will be recorded for all patients.

Experimental Design Aim 2: The computer-based simulation of CAS is performed exploiting a computational framework, which can be used to analyze both stent apposition and vessel wall stress in a virtual manner. The framework accounts for two main parts: the vessel model and stent model. Preoperative and postoperative medical images (including high resolution Contrast Enhanced (CE)-MRI and Computed Tomography Angiography (CTA)) will represent the input to build a patient specific carotid model. The 3D lumen profile of the vessel is reconstructed through the segmentation of DICOM image stack using tools like ITK-SNAP (www.itksnap.org) or VMTK (www.vmtk.org). The computational domain (the so-called mesh), used to solve the equilibrium equations governing the structural stent-vessel interaction, is created by an in-house developed procedure, coded in Matlab (The Mathworks Inc., Natick,MA, USA). The non-linear mechanical response of the arterial tissue is reproduced adopting an anisotropic hyperelastic strain-energy function, accounting for two families of fibers, oriented along a preferred direction with a certain degree of dispersion. The model parameters will be calibrated with respect to experimental tensile tests of the carotid tissue. The arterial model is then assembled in the simulation environment with a given stent model, picked from a predefined library of stent designs (the stent mesh generation is based on geometrical measurements performed on high-resolution micro-CT of stent samples). The CAS simulation is performed through structural finite element analysis (FEA); the commercial FEA solver Abaqus (Simulia, Dassault Systemes, FR), is adopted to run the simulations. The engineering outcomes of the simulations, (i.e. the nodal displacement field, stress tensor and strain at each integration points of the mesh), are elaborated to assess clinically relevant parameters of stenting performance (e.g. lumen gain, vessel straightening, stent cell size). The output will be used as an input of the Computational Fluid Dynamics analysis to evaluate the impact of the implanted design on the local haemodynamics (e.g., wall shear stress, oscillatory shear index, etc). Similarly, the structural analysis of CEA will be performed through the virtual pressurization of the post-operative arterial geometry.

Experimental design 3: Moving from Computational Fluid Dynamics and Fluid-Structure Interaction analysis, the investigators plan to introduce a specific model to describe the baroreflex function and this may be affected by the two different types of treatment (CEA and CAS). This requires the set up of a so-called "geometrical multiscale" model. With this, the investigators mean a numerical model coupling a local description of the hemodynamics (the one developed in Aim 2) with a more systemic representation. The latter consists of two components:

a) a 1D network mathematically described by a system of partial differential equations representing the propagation of the pressure wave along the arterial tree; each segment of the network is given by a hyperbolic system called "Euler equations" b) a compartment model for representing the peripheral microcirculation and for including the feedback mechanisms induced by the baroreflex function. Following, this will be represented by a system of ordinary differential equations where resistances properly depend on the baroreflex function.

In this aim the investigators plan two sub-aims:

1. Set up of a computational multiscale model within the framework of the LifeV solver, a finite element general purpose C++ Object Oriented library, developed by A. Veneziani and his collaborators (in Milan Politecnico and Lausanne EPFL) www.lifev.org and openly downloadable. At this stage, the investigators will reproduce the general model of Blanco et al. In particular, the identification of the parameters for the two different levels of models (1D and Lumped Parameters) will be carried out following the procedure suggested. Validation of the solver will also take advantage of the benchmarks presented in this paper.
2. Adoption of the solver previously developed for the test cases considered in Aim 2. This means that the 3D model developed in Aim 2 will be adopted for the 3D part of the geometrical multiscale model. This will allow to provide a quantitative analysis of the different impact of the two treatments and ultimately to assess in a virtual scenario how the changes of carotid compliance may impair the baroreflex function. All the CAS and CEA cases considered in Aim 2 will be equipped of this multiscale framework. The expected deliverables of this aim are therefore: a) a validated open source geometrical multiscale solver including the baroreflex function to be used systematically in patient-specific settings. b) extensive comparison of the performances of the different options.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patients with >=70% symptomatic or >=80% asymptomatic internal carotid stenosis

Exclusion Criteria:

* Incapability to give informed consent
* Previous disabling stroke
* Contralateral carotid occlusion or >70% stenosis
* Systemic disease judged non compatible with the procedures or randomization
* Suspected or manifested pregnancy
* General contraindications to MRI or CT studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
R-R interval (sec) and Systolic Arterial Pressure (SAP) (mmHg) in rest and tilt position for baroreceptor function | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA

SECONDARY OUTCOMES:
Cognitive P300 latency (ms) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Mean and maximum flow velocity magnitude (cm/sec) in common carotid artery (CCA) and internal carotid artery (ICA) along the cardiac cycle | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Systolic wall shear stress (dyn/cm2) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Time-averaged wall shear stress (TAWSS) (dyn/cm2) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Oscillatory index (OSI) (%) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Flow helicity (-) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
CCA/ICA Flow split (%) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Common carotid artery (CCA) - internal carotid artery (ICA) mean and maximum pressure drop (mmHg) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Carotid wall von Mises stress (dyn/cm2) at the systolic peak | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Carotid wall maximum principal stress (dyn/cm2) at the systolic peak and corresponding directions (-) Maximum, mean, and min principal strain (-) and corresponding directions (-) | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Carotid augmentation index (%) of pressure wave | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA
Effective reflecting distance (mm) of pressure wave | 20 months
  Comparison pre- and post-CAS, Comparison pre- and post-CEA

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutlip DE, Pinto DS. Extracranial carotid disease revascularization. Circulation. 2012 Nov 27;126(22):2636-44. doi: 10.1161/CIRCULATIONAHA.112.110411. No abstract available. PMID 23184283
- [Background] Marrocco-Trischitta MM, Cremona G, Lucini D, Natali-Sora MG, Cursi M, Cianflone D, Pagani M, Chiesa R. Peripheral baroreflex and chemoreflex function after eversion carotid endarterectomy. J Vasc Surg. 2013 Jul;58(1):136-44.e1. doi: 10.1016/j.jvs.2012.11.130. Epub 2013 Apr 28. PMID 23632295
- [Background] Hayase H, Tokunaga K, Nakayama T, Sugiu K, Nishida A, Arimitsu S, Hishikawa T, Ono S, Ohta M, Date I. Computational fluid dynamics of carotid arteries after carotid endarterectomy or carotid artery stenting based on postoperative patient-specific computed tomography angiography and ultrasound flow data. Neurosurgery. 2011 Apr;68(4):1096-101; discussion 1101. doi: 10.1227/NEU.0b013e318208f1a0. PMID 21221041
- [Background] Irvine CD, Gardner FV, Davies AH, Lamont PM. Cognitive testing in patients undergoing carotid endarterectomy. Eur J Vasc Endovasc Surg. 1998 Mar;15(3):195-204. doi: 10.1016/s1078-5884(98)80176-7. PMID 9587331
- [Background] Bohm M, Cotton D, Foster L, Custodis F, Laufs U, Sacco R, Bath PM, Yusuf S, Diener HC. Impact of resting heart rate on mortality, disability and cognitive decline in patients after ischaemic stroke. Eur Heart J. 2012 Nov;33(22):2804-12. doi: 10.1093/eurheartj/ehs250. Epub 2012 Aug 26. PMID 22922507
- [Background] Davies PF. Overview: temporal and spatial relationships in shear stress-mediated endothelial signalling. J Vasc Res. 1997 May-Jun;34(3):208-11. doi: 10.1159/000159224. No abstract available. PMID 9226302
- [Background] Hathcock JJ. Flow effects on coagulation and thrombosis. Arterioscler Thromb Vasc Biol. 2006 Aug;26(8):1729-37. doi: 10.1161/01.ATV.0000229658.76797.30. Epub 2006 Jun 1. PMID 16741150
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Auricchio F, Conti M, De Beule M, De Santis G, Verhegghe B. Carotid artery stenting simulation: from patient-specific images to finite element analysis. Med Eng Phys. 2011 Apr;33(3):281-9. doi: 10.1016/j.medengphy.2010.10.011. Epub 2010 Nov 9. PMID 21067964
- [Background] Conti M, Van Loo D, Auricchio F, De Beule M, De Santis G, Verhegghe B, Pirrelli S, Odero A. Impact of carotid stent cell design on vessel scaffolding: a case study comparing experimental investigation and numerical simulations. J Endovasc Ther. 2011 Jun;18(3):397-406. doi: 10.1583/10-3338.1. PMID 21679082
- [Background] Auricchio F, Conti M, Ferrara A, Morganti S, Reali A. Patient-specific finite element analysis of carotid artery stenting: a focus on vessel modeling. Int J Numer Method Biomed Eng. 2013 Jun;29(6):645-64. doi: 10.1002/cnm.2511. Epub 2012 Sep 29. PMID 23729192
- [Background] Auricchio F, Conti M, Ferraro M, Reali A. Evaluation of carotid stent scaffolding through patient-specific finite element analysis. Int J Numer Method Biomed Eng. 2012 Oct;28(10):1043-55. doi: 10.1002/cnm.2509. Epub 2012 Aug 25. PMID 23027634
- [Background] De Santis G, Conti M, Trachet B, De Schryver T, De Beule M, Degroote J, Vierendeels J, Auricchio F, Segers P, Verdonck P, Verhegghe B. Haemodynamic impact of stent-vessel (mal)apposition following carotid artery stenting: mind the gaps! Comput Methods Biomech Biomed Engin. 2013;16(6):648-59. doi: 10.1080/10255842.2011.629997. Epub 2011 Dec 8. PMID 22149183
- [Background] De Santis G, Trachet B, Conti M, De Beule M, Morbiducci U, Mortier P, Segers P, Verdonck P, Verhegghe B. A computational study of the hemodynamic impact of open- versus closed-cell stent design in carotid artery stenting. Artif Organs. 2013 Jul;37(7):E96-106. doi: 10.1111/aor.12046. Epub 2013 Apr 12. PMID 23578331
- [Background] Blanco PJ, Trenhago PR, Fernandes LG, Feijoo RA. On the integration of the baroreflex control mechanism in a heterogeneous model of the cardiovascular system. Int J Numer Method Biomed Eng. 2012 Apr;28(4):412-33. doi: 10.1002/cnm.1474. Epub 2011 Nov 2. PMID 25365656
- [Background] Towfighi A, Saver JL. Stroke declines from third to fourth leading cause of death in the United States: historical perspective and challenges ahead. Stroke. 2011 Aug;42(8):2351-5. doi: 10.1161/STROKEAHA.111.621904. Epub 2011 Jul 21. PMID 21778445
- [Background] Bunch CT, Kresowik TF. Can randomized trial outcomes for carotid endarterectomy be achieved in community-wide practice? Semin Vasc Surg. 2004 Sep;17(3):209-13. doi: 10.1016/s0895-7967(04)00043-2. PMID 15449242